CLINICAL TRIAL: NCT02256787
Title: Safety, Tolerance, and Pharmacokinetics of Single Oral Doses of 5 mg, 20 mg, 60 mg, 120 mg, 200 mg, 300 mg, 600 mg, 1000 mg, 1500 mg, 2000 mg, 2400 mg, and 3000 mg BILB 1941 ZW (PEG 400/TRIS Solution) in Healthy Male Subjects, in a Randomised Double Blind, Placebo Controlled Rising Dose Study, Followed With an Open-label Intra-subject Three-Way Crossover Bioavailability Comparison of 600 mg BILB 1941 ZW in a PEG 400/TRIS Solution and 600 mg BILB 1941 ZW Tablet and 600 mg BILB 1941 ZW Tablet Administered With Food
Brief Title: Safety, Tolerance, and Pharmacokinetics of Single Rising Oral Doses of BILB 1941 ZW Solution in Healthy Male Subjects, Followed With Bioavailability Comparison of BILB 1941 ZW Tablet and Solution Formulation Administered With or Without Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1201.1
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (5):
- BILB 1941 ZW - single rising dose (Experimental): Single rising dose part
  Interventions: Drug: BILB 1941 ZW - single rising dose part
- Placebo (Placebo Comparator): Single rising dose part
  Interventions: Drug: Placebo
- BILB 1941 ZW - tablet - fasted (Experimental): Relative bioavailability: The oral solution fasted should be compared with the solid form fasted and after a standardized breakfast
  Interventions: Drug: BILB 1941 ZW - tablet
- BILB 1941 ZW - solution (Experimental): Relative bioavailability: The oral solution fasted should be compared with the solid form fasted and after a standardized breakfast
  Interventions: Drug: BILB 1941 ZW - solution
- BILB 1941 ZW - tablet - fed (Experimental): Relative bioavailability: The oral solution fasted should be compared with the solid form fasted and after a standardized breakfast
  Interventions: Drug: BILB 1941 ZW - tablet; Other: standardized breakfast

INTERVENTIONS:
Drug: BILB 1941 ZW - single rising dose part
  Arms: BILB 1941 ZW - single rising dose
Drug: Placebo
  Arms: Placebo
Drug: BILB 1941 ZW - solution
  Arms: BILB 1941 ZW - solution
Drug: BILB 1941 ZW - tablet
  Arms: BILB 1941 ZW - tablet - fasted; BILB 1941 ZW - tablet - fed
Other: standardized breakfast
  Arms: BILB 1941 ZW - tablet - fed

SUMMARY:
The objective of the current study was to investigate the safety, tolerability, and pharmacokinetics of BILB 1941 ZW following the administration of single rising doses from 5 mg to 300 mg. In addition the bioavailability of the 60 mg dose given fasted and after a high-fat breakfast was to be be investigated

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males according to the following criteria based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests:

   1.1 No finding deviating from normal and of clinical relevance

   1.2 No evidence of a clinically relevant concomitant disease
2. Age ≥18 and Age ≤50 years, BMI ≥18.5 and BMI ≤29.9 kg/m2 (Body Mass Index)
3. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* History or current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders, including a clinical history of viral hepatitis, or serological evidence of active Hepatitis B or Hepatitis C infection
* History of orthostatic hypotension, fainting spells and blackouts
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within 1 month prior to administration
* Use of any drugs which might influence the results of the trial within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within 1 month prior to administration or during the trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation of more than 100 mL within 1 month prior to administration or during the trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Any laboratory value outside the clinically accepted reference range and of clinical relevance
* History of any familial bleeding disorder

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2004-01; Primary Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects with abnormal findings in physical examination | up to 48 hours following drug administration
Number of subjects with abnormal changes in laboratory parameters | up to 48 hours following drug administration
Number of subjects with clinically significant changes in vital signs | up to 48 hours following drug administration
  Blood pressure, Pulse Rate
Number of subjects with adverse events | up to 48 hours following drug administration
Number of subjects with clinically significant changes in 12-lead ECG (electrocardiogram) | up to 48 hours following drug administration
Assessment of tolerability by investigator on a 4-point scale | after 48 hours following drug administration

SECONDARY OUTCOMES:
Cmax (maximum concentration of the analyte in plasma) | up to 48 hours following drug administration
tmax (time from dosing to maximum concentration) | up to 48 hours following drug administration
AUC0-∞ (area under the concentration time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 48 hours following drug administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) | up to 48 hours following drug administration
λz (terminal rate constant in plasma) | up to 48 hours following drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 48 hours following drug administration
MRT (Mean time of residence of drug molecules in the body after intravascular administration) | up to 48 hours following drug administration
Vz/F (Apparent volume of distribution during the terminal phase after extravascular administration) | up to 48 hours following drug administration